CLINICAL TRIAL: NCT03436745
Title: A Pilot Study to Evaluate the Effects of Castration on the Pharmacokinetics of Zolpidem After Single Dose Administration in Men With Prostate Cancer Undergoing Androgen Deprivation Therapy Compared to Normal Healthy Females
Brief Title: The Effects of Castration on the Pharmacokinetics of Zolpidem After Single Dose Administration In Men With Prostate Cancer Undergoing Androgen Deprivation Therapy Compared to Normal Healthy Females
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Figg, Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 180058; 18-C-0058
Record Dates: First submitted 2018-02-16; First posted 2018-02-19 (Actual); Results first posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Prostatic Neoplasms
Keywords: Insomnia; Enzyme Expression; PSA; TESTOSTERONE; Recommended Dose
MeSH Terms: conditions — Prostatic Neoplasms; Sleep Initiation and Maintenance Disorders | interventions — Zolpidem; Electrocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Female (Active Comparator): Single 5 mg oral dose of zolpidem
  Interventions: Drug: Zolpidem; Diagnostic Test: ECG
- Zolpidem pre and post castration (Experimental): 5 mg oral dose of zolpidem prior to undergoing androgen deprivation therapy (ADT) followed by 5 mg oral dose of zolpidem after ADT and testosterone reaches castrate levels
  Interventions: Drug: Zolpidem; Diagnostic Test: ECG

INTERVENTIONS:
Drug: Zolpidem — In men with prostate cancer, males (pre-castration, n=8-10) will receive oral zolpidem in the form of a 5 mg tablet. Blood samples will be collected for pharmacokinetic analysis at pre-dose and 0.5, 1, 2, 4, and 8-hours post-dose. This cohort of men will then undergo androgen deprivation therapy with standard doses of goserelin. When castrate testosterone levels reach <50 ng/dL (post-castration), they will receive another 5 mg single dose of zolpidem followed by 8-hr pharmacokinetic (PK) evaluation of zolpidem and its metabolites. Normal healthy females (n=5-8) will receive treatment with a single dose of 5 mg tablet of zolpidem followed by 8-hr PK evaluation of zolpidem and its metabolites. Blood samples will be collected for PK analysis at pre-dose and 0.5, 1, 2, 4, and 8-hours post-dose.
  Other Names: Ambien; Zolpimist; Edluar
Diagnostic Test: ECG — Screening and baseline.
  Other Names: Electrocardiogram

SUMMARY:
Background:

Insomnia is associated with difficulty sleeping. The drug zolpidem is widely prescribed for insomnia. Women have reported worse effects from the drug than men. Women have higher amounts of zolpidem in their body that may persist after waking. Drug exposure may also depend on male hormones that change during prostate cancer therapy. Researchers want to see if these findings can provide a more-accurate dose to healthy women and men with prostate cancer.

Objective:

To study amounts of zolpidem in men who have been diagnosed with prostate cancer before they are castrated and after, and to compare these results to healthy women s.

Eligibility:

Men ages 18 and older who have been diagnosed with prostate cancer who are planning to receive androgen deprivation therapy (ADT)

Healthy women age 18 and older

Design:

Participants will be screened with:

Blood tests

Physical exam

Electrocardiogram (EKG) heart test

Male participants will confirm their prostate cancer. This can be done with a tumor sample tissue from a previous surgery or a report from a doctor.

Female participants may have a pregnancy test.

Participants will be admitted to the clinic in the evening and stay overnight. They will:

Take a 5 mg zolpidem tablet on an empty stomach around 11 p.m.

Have blood drawn multiple times

Have physical exams and EKGs

Answer questions about their symptoms and medicines they are taking

Male participants will have ADT as part of their standard cancer treatment. After that, the testosterone in their blood will be measured. They will repeat the overnight clinic stay.

Participants will get a follow-up phone call after each stay.

DETAILED DESCRIPTION:
Background:

* Zolpidem is currently approved for the treatment of patients with insomnia.
* Women reported experiencing an increased incidence of adverse effects than men, resulting in a reduction of the recommended dose of zolpidem for women.
* Zolpidem metabolism is affected by both age and gender; the recommended dose for the elderly and female populations is 5mg daily.
* Subsequent studies have shown that women experience greater exposure to zolpidem than men, potentially due to androgen-driven differences in enzyme expression.
* A preclinical study showed that castrated male rats exhibited zolpidem pharmacokinetics similar to that of female rats, providing further evidence to suggest that zolpidem pharmacokinetics are androgen-driven.

Objectives:

-To evaluate the effect of castration on the pharmacokinetics of a single 5-mg dose of zolpidem in participants with prostate cancer undergoing androgen deprivation therapy (previous post-castration therapy) compared to normal healthy females.

Eligibility:

* Participants with prostate cancer (rising prostate-specific antigen (PSA) and greater than or equal to 100 ng/dL)
* Females in good health condition or without significant diseases
* After androgen deprivation therapy, castrate testosterone levels <50 ng/dL
* Eastern Cooperative Oncology Group (ECOG) 0-1

Design:

* Comparative, single-dose pharmacokinetic study.
* Men with prostate cancer (pre-castration) and normal healthy females will receive treatment with a single dose of 5 mg tablet of zolpidem followed by 8-hour pharmacokinetic evaluation of zolpidem and its metabolites.
* Men will then undergo androgen deprivation therapy and when castrate testosterone levels <50 ng/dL (post-castration), they will receive another 5 mg single dose of zolpidem followed by 8-hour pharmacokinetic evaluation of zolpidem and its metabolites.
* Normal healthy females will receive treatment with a single dose of 5 mg tablet of zolpidem followed by 8-hour pharmacokinetic evaluation of zolpidem and its metabolites.

ELIGIBILITY:
* INCLUSION CRITERIA - FOR MALE COHORT:
* Patients must have histologically or cytologically confirmed prostate cancer. Note: If histologic documentation is unavailable, a clinical course consistent with prostate cancer is acceptable.
* Patients must be eligible for and must be planning to undergo androgen deprivation therapy
* Testosterone levels greater than or equal to 100 ng/dL
* Patients must have progressive prostate cancer as indicated by either prostate-specific antigen (PSA) progression (PSA progression is defined as two consecutively rising PSAs above the nadir post- definitive therapy and an absolute value greater than 1.0 ng/mL separated by at least 2 weeks) or radiographic progression based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Prostate Cancer Working Group 3 (PCWG3).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Patients must have normal organ and marrow function as defined below:

  * Hemoglobin greater than or equal to 9 g/dL
  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 150,000/mcL
  * total bilirubin within normal institutional limits
  * Aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) serum glutamic-pyruvic transaminase (SGPT) less than or equal to institutional upper limit of normal
  * creatinine within normal institutional limits OR creatinine clearance greater than or equal to 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (calculated via Cockcroft-Gault equation)
* Patients must not have other concurrent malignancies (within the past 2 years with the exception of non-melanoma skin cancer and Rai Stage 0 chronic lymphocytic leukemia), in situ carcinoma of any site, or life-threatening illnesses, including untreated infection (must be at least 1 week off intravenous antibiotic therapy before beginning zolpidem).
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Ability to swallow study medication.
* Willingness to travel to National Institutes of Health (NIH) for follow-up visits.
* Men age greater than or equal to 18 years of age. Children are excluded because prostate cancer is not common in pediatric populations.

INCLUSION CRITERIA - FOR NORMAL HEALTHY FEMALE COHORT:

* Females age greater than or equal to 18 years of age
* Good health conditions or without significant diseases, according to best medical judgement.
* If breastfeeding, must be willing to discard breastmilk for 24 hours following zolpidem.
* Ability if subject to understand and the willingness to sign a written informed consent Ability to swallow study medication.

EXCLUSION CRITERIA - FOR MALE COHORT:

* Patients who are receiving any other investigational agents (in the past 28 days) or herbal medications (within 1 day).
* Patients who have received systemic chemotherapy for prostate cancer will not be eligible.
* Known hypersensitivity to Zolpidem or chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug.
* Clinically significant cardiac disease, e.g. New York Heart Association (NYHA) classes III-IV; uncontrolled angina, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction in the previous 6 months as confirmed by an electrocardiogram (ECG).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with zolpidem. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with known active treatment for Hepatitis B and C infections.
* Patients who are taking medications that may alter the metabolism of zolpidem. This includes strong Cytochrome P450 3A4 (CYP3A4) inhibitors or inducers or CYP3A4 substrates with a narrow therapeutic index. For a current table of Substrates, Inhibitors and Inducers please access the following website: http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm
* History or presence of hepatic or gastrointestinal diseases, or other condition that interferes with drug absorption, distribution, excretion or metabolism.
* Patients currently taking other sedative hypnotic medications Patients with a known history of psychiatric issues
* Patients at risk for fall or who have had recent fractures
* Patients of Asian descent

EXCLUSION CRITERIA - FOR NORMAL HEALTHY FEMALE COHORT:

* Chronic therapy with any drugs, except contraceptives
* History of hepatic, kidney, lungs, gastrointestinal, epileptic, hematologic or psychiatric disease; hypotension or hypertension, of any etiology, that requires pharmacological treatment; history of myocardial infarction, angina and/or heart failure.
* Use of regular medications within 2 weeks prior study enrollment or use of any medications within one week prior to study enrollment, except contraceptives or cases which, based on drugs or metabolites half-life, complete elimination can be assumed.
* Hospitalization for any reason up to 8 weeks before enrollment.
* Any condition, according to investigator's best judgement, that prevents the subject to participate in the trial
* Pregnancy, labor or miscarriage within 12 weeks before admission predicted date.
* Known hypersensitivity to zolpidem or chemically related compounds; history of serious adverse reactions or hypersensitivity to any drug.

Females of Asian descent

-History of taking estrogen derivatives, androgens, or similar hormonal replacement or supplementation products. Past and current use of hormonal contraceptives is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-C-0058.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Female Cohort: One Time Zolpidem: Single 5 mg oral dose of zolpidem Dose Level 2 Zolpidem: In men with prostate cancer, males (pre-castration, n=8-10) will receive oral zolpidem in the form of a 5 mg tablet. Blood samples will be collected for pharmacokinetic analysis at pre-dose and 0.5, 1, 2, 4, and 8-hours post-dose. This cohort of men will then undergo androgen deprivation therapy with standard doses of goserelin. When castrate testosterone levels reach <50 ng/dL (post-castration), they will receive another 5 mg single dose of zolpidem followed by 8-hr pharmacokinetic (PK) evaluation of zolpidem and its metabolites. Normal healthy females (n=5-8) will receive treatment with a single dose of 5 mg tablet of zolpidem followed by 8-hr PK evaluation of zolpidem and its metabolites. Blood samples will be collected for PK analysis at pre-dose and 0.5, 1, 2, 4, and 8-hours post-dose.
- Prostate Cancer Cohort: Zolpidem Pre and Post Castration: 5 mg oral dose of zolpidem prior to undergoing androgen deprivation therapy (ADT) followed by 5 mg oral dose of zolpidem after ADT and testosterone reaches castrate levels Dose Level 1a -> Dose Level 1b. Zolpidem: In men with prostate cancer, males (pre-castration, n=8-10) will receive oral zolpidem in the form of a 5 mg tablet. Blood samples will be collected for pharmacokinetic analysis at pre-dose and 0.5, 1, 2, 4, and 8-hours post-dose. This cohort of men will then undergo androgen deprivation therapy with standard doses of goserelin. When castrate testosterone levels reach <50 ng/dL (post-castration), they will receive another 5 mg single dose of zolpidem followed by 8-hr pharmacokinetic (PK) evaluation of zolpidem and its metabolites. Normal healthy females (n=5-8) will receive treatment with a single dose of 5 mg tablet of zolpidem followed by 8-hr PK evaluation of zolpidem and its metabolites. Blood samples will be collected for PK analysis at pre-dose and 0.5, 1, 2, 4, and 8-hours post-dose.
- Enrolled But Not Treated: Participant was enrolled but not treated.
Period: Overall Study
Arm/Group | Healthy Female Cohort: One Time Zolpidem | Prostate Cancer Cohort: Zolpidem Pre and Post Castration | Enrolled But Not Treated
Started | 10 | 1 | 1
Follow-up Period Completed | 10 | 1 | 0
Completed | 10 | 1 | 0
Not Completed | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were collected for one participant enrolled and not treated and is reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Cancer Cohort: Zolpidem Pre and Post Castration | Healthy Female Cohort: One Time Zolpidem | Enrolled But Not Treated | Total
Number analyzed (Participants) | 1 | 10 | 1 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 10 | 0 | 11
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (0) | 27.6 (4.2) | 75 (0) | 34.58 (16.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 10 | 0 | 10
  Male | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 0 | 3
  Not Hispanic or Latino | 1 | 7 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 6 | 0 | 6
  White | 1 | 4 | 1 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 10 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Area Under the Plasma Concentration 0-8Hour (Hr)(AUC0-8hr) Values in Males Between Pre-Androgen Deprivation Therapy (ADT) and Post-ADT
Description: AUC is a measure of the serum concentration of Zolpidem over time. It is used to characterize drug absorption. The AUC values will be compared between the time points for males to see if the AUC increases significantly. Pre-ADT males will be subtracted from the paired values in males once they are post-ADT and tested for a difference using a paired t-test with a two-sided 0.05 significance level, or a Wilcoxon signed rank test if the paired differences are not normally distributed.
Time Frame: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, and 8-hours post-dose.
Measure: Mean (95% Confidence Interval); unit: Hr*ng/mL
Groups:
- Prostate Cancer Cohort: Zolpidem Pre-Castration: Zolpidem: In men with prostate cancer, males (pre-castration) will receive oral zolpidem in the form of a 5 mg tablet.
- Prostate Cancer Cohort: Zolpidem Post Castration: This cohort of men will undergo androgen deprivation therapy with standard doses of goserelin. When castrate testosterone levels reach <50 ng/dL (post-castration), they will receive another 5 mg single dose of zolpidem.
Arm/Group | Prostate Cancer Cohort: Zolpidem Pre-Castration | Prostate Cancer Cohort: Zolpidem Post Castration
Number analyzed (Participants) | 1 | 1
Hr*ng/mL | 484.65 [NA to NA] — 95% confidence interval cannot be calculated because we only have 1 male enrolled, so we cannot scientifically make a comparison. | 473.05 [NA to NA] — 95% confidence interval cannot be calculated because we only have 1 male enrolled, so we cannot scientifically make a comparison.

2. Secondary Outcome: Comparison of Area Under the Plasma Concentration 0-8Hour (Hr)(AUC0-8hr) Values Between Post-Androgen Deprivation Therapy (ADT) Males and Healthy Female Participants
Description: AUC is a measure of the serum concentration of Zolpidem over time. It is used to characterize drug absorption. AUC values will be compared between those of post-ADT males and healthy females to assess whether AUC values are approximately equivalent between post-ADT males and healthy females.
Time Frame: pre-dose and 0.25, 0.5, 1, 1.5, 2, 3, 4, and 8-hours post-dose.
Measure: Mean (90% Confidence Interval); unit: Hr*ng/mL
Groups:
- Healthy Female Cohort: One Time Zolpidem: Normal healthy females will receive treatment with a single dose of 5 mg tablet of zolpidem.
Arm/Group | Healthy Female Cohort: One Time Zolpidem | Prostate Cancer Cohort: Zolpidem Post Castration
Number analyzed (Participants) | 10 | 1
Hr*ng/mL | 242 [7.2 to 478.05] | 473.05 [NA to NA] — 95% confidence interval cannot be calculated because we only have 1 male enrolled, so we cannot scientifically make a comparison.

3. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0).
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Study Period 1, Day 1 to Day 3 (female &male cohort). From first intervention, Study Period Day 1 to 3 days after removal from study treatment, approximately 3 days. Study Period 2, Day 1 to Day 3 (male cohort) after removal from study treatment, =3 days.
Measure: Count of Participants; unit: Participants
Groups:
- Prostate Cancer Cohort: Zolpidem Pre and Post Castration: 5 mg oral dose of zolpidem prior to undergoing androgen deprivation therapy (ADT) followed by 5 mg oral dose of zolpidem after ADT and testosterone reaches castrate levels
  Zolpidem: In men with prostate cancer, males (pre-castration) will receive oral zolpidem in the form of a 5 mg tablet. This cohort of men will then undergo androgen deprivation therapy with standard doses of goserelin. When castrate testosterone levels reach <50 ng/dL (post-castration), they will receive another 5 mg single dose of zolpidem.
Arm/Group | Healthy Female Cohort: One Time Zolpidem | Prostate Cancer Cohort: Zolpidem Pre and Post Castration
Number analyzed (Participants) | 10 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Study Period 1, Day 1 to Day 3 (female &male cohort). From first intervention, Study Period Day 1 to 3 days after removal from study treatment, approximately 3 days. Study Period 2, Day 1 to Day 3 (male cohort) after removal from study treatment, =3 days.
Groups:
- Healthy Female Cohort: One Time Zolpidem: Normal healthy females (n=5-8) will receive treatment with a single dose of 5 mg tablet of zolpidem.
Arm/Group | Healthy Female Cohort: One Time Zolpidem | Prostate Cancer Cohort: Zolpidem Pre and Post Castration
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/1
Other Adverse Events (participants affected / at risk) | 1/10 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Female Cohort: One Time Zolpidem (N=10) | Prostate Cancer Cohort: Zolpidem Pre and Post Castration (N=1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT03436745/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/45/NCT03436745/ICF_001.pdf